CLINICAL TRIAL: NCT04780412
Title: Efficacy of Misoprostol in Prevention of Neonatal Respiratory Morbidity in Parturient at Early Term Elective Caesarian Section
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Samar Ali, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Misoprostol
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Transient Tachypnea of the Newborn; Neonatal Respiratory Distress
MeSH Terms: conditions — Transient Tachypnea of the Newborn; Pulmonary Atelectasis | interventions — Misoprostol; Alprostadil

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol Group (Active Comparator)
  Interventions: Drug: Misoprostol
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — Vaginal Misoprostol tablets in a dose of 50 microgram given 90-120 minutes before an elective caesarian section.
  Other Names: prostaglandin E1
  Arms: Misoprostol Group
Drug: Placebo — Vaginal placebo pills given 90-120 minutes before an elective caesarian section.
  Arms: Placebo Group

SUMMARY:
Neonatal respiratory morbidities represent a common group of post natal complications including respiratory distress syndrome, transient tachypnea of newborn, and persistent pulmonary hypertension of newborn.

It is thought that preoperative vaginal misoprostol administration may decrease the incidence of neonatal respiratory morbidity especially transient tachypnea of newborn. And therefore, it may decrease the incidence of admission to neonatal intensive care units for respiratory causes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or more.
* Early term singleton pregnancy.
* Elective caesarian section at (37 - 38+6) weeks of gestation.
* Any indication for lower uterine segment caesarian section other than labor (as malpresentations, severe preeclampsia, placenta previa with no previous bleeding attacks, Diabetes Mellitus, macrosomic fetus, non reassuring cardiotocogram (CTG), and fetal growth restriction).
* Informed written consent signed by the participating pregnant woman.

Exclusion Criteria:

* Women having any contraindication to Prostaglandin E1 as hypersensitivity, respiratory disease (especially bronchial asthma), or glaucoma.
* Any mental problems that block understanding of the nature and all the possible consequences of the procedure and the study.
* Pregnancies of known fetal diseases or chromosomal abnormalities.
* Non-singleton pregnancies.
* Emergency caesarian section as in ruptured membrane and women in labor pain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
incidence of neonatal respiratory morbidity (NRM) | up to 24 hours after birth
  The incidence of neonatal respiratory morbidity, especially transient tachypnea of newborn, in early term neonates born to elective caesarian section.

SECONDARY OUTCOMES:
Neonatal intensive care unit (NICU) admission | up to 24 hours after birth
  The incidence of the need for neonatal intensive care unit admission during the first ten days after delivery in early term neonates born to elective caesarian section.

CONTACTS AND LOCATIONS:
Overall Officials: Samar A. Kandeel, Principal Investigator — Ain Shams University - Faculty of Medicine
Locations (1):
- Ain Shams University - Faculty of Medicine, Cairo, Egypt